CLINICAL TRIAL: NCT06082583
Title: A Randomized Controlled Trial of the Efficacy of Combining Traditional Tibetan and Remote Ischemic Conditioning on High Altitude Polycythemia
Brief Title: The Efficacy of Combination of Traditional Tibetan and Remote Ischemic Conditioning on High Altitude Polycythemia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HAPC
Record Dates: First submitted 2023-09-21; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: High Altitude Polycythemia
MeSH Terms: interventions — Medicine, Tibetan Traditional

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tibetan Medicine Group (Active Comparator)
  Interventions: Drug: Tibetan Medicine (Shiliu Jianwei Powder, Ershiwuwei Yuganzi Pills, Qiwei Tiexue Pill)
- Tibetan Medicine-Remote Ischemic Conditioning Group (Experimental)
  Interventions: Device: Remote Ischemic Conditioning; Drug: Tibetan Medicine (Shiliu Jianwei Powder, Ershiwuwei Yuganzi Pills, Qiwei Tiexue Pill)

INTERVENTIONS:
Device: Remote Ischemic Conditioning — Remote ischemic conditioning conducted by an electric auto-control device will be performed twice a day for 14 days, each session including 5-min ischemia and 5-min reperfusion.
  Other Names: An electric auto-control device to perform remote ischemic conditioning.
  Arms: Tibetan Medicine-Remote Ischemic Conditioning Group
Drug: Tibetan Medicine (Shiliu Jianwei Powder, Ershiwuwei Yuganzi Pills, Qiwei Tiexue Pill) — Comprehensively Tibetan medicine for 28 days, including Shiliu Jianwei Powder, Ershiwuwei Yuganzi Pills and Qiwei Tiexue Pill, dosage of which are 1.5g daily.

SUMMARY:
A multicenter, randomized controlled trial was designed to evaluate the effectiveness and safety of the comprehensive traditional Tibetan medicine program combined with remote ischemic conditioning on high altitude polycythemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high-altitude polycythemia aging 18 to 65 years.

Exclusion Criteria:

* Allergic to Tibetan medicine ingredients;
* Inappropriate to receive Tibetan medicine treatment and/or remote ischemic conditioning.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of effective treatment | Baseline and 1 month after treatment.
  The hemoglobin levels decreased ≥20% after treatment compared to pre-treatment.

IPD SHARING:
Plan to Share IPD: No